CLINICAL TRIAL: NCT03560167
Title: An Early Feasibility Study of the AccuCinch® Ventricular Restoration System in Patients With Prior Mitral Valve Intervention (PMVI) and Recurrent Mitral Regurgitation - The CorCinch-PMVI Study
Brief Title: Early Feasibility Study of the AccuCinch® Ventricular Restoration System in Patients With Prior Mitral Valve Intervention (PMVI) and Recurrent Mitral Regurgitation
Acronym: CorCinch-PMVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ancora Heart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 5018
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure; Cardiomyopathy, Dilated
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AccuCinch® Ventricular Restoration System (Experimental)
  Interventions: Device: AccuCinch® Ventricular Restoration System

INTERVENTIONS:
Device: AccuCinch® Ventricular Restoration System — AccuCinch® Ventricular Restoration System in Patients with Prior Mitral Valve Intervention (PMVI) and Recurrent Mitral Regurgitation

SUMMARY:
This is a non-randomized, prospective, multi-center Early Feasibility Study of the AccuCinch® Ventricular Restoration System in Patients with Prior Mitral Valve Intervention (PMVI) and Recurrent Mitral Regurgitation.

DETAILED DESCRIPTION:
Device name changed from AccuCinch® Ventricular Repair System to AccuCinch® Ventricular Restoration System, FDA Approval Date August 14, 2020.

ELIGIBILITY:
Inclusion Criteria:

* Study patient is at least 18-years old
* Severity of FMR: ≥ Moderate (i.e., ≥2+, according to Stone et al Clinical Trial Design Principles and Endpoint Definitions for Transcatheter Mitral Valve Repair and Replacement: Part 1: Clinical Trial Design Principles. A Consensus Document from the Mitral Valve Academic Research Consortium1; and 2003 ASE Guidelines for grading mitral regurgitation2)
* Patient has had a prior surgical or percutaneous mitral repair procedure >3 months prior to enrollment
* LV Ejection Fraction: ≥20 to ≤40%
* Symptom Status: NYHA II-IV (i.e., ambulatory)
* Prescribed appropriate guideline-directed medical therapy for heart failure for at least 3 months with stable doses of diuretics, beta-blockers and Angiotensin converting enzyme inhibitor (ACEi) or Angiotensin II Receptor Blockers (ARB) for 1 month (with stable defined as no greater than 100% increase of 50% decrease in medication doses). Treatment shall include CRT and/or ICD when indicated by guidelines.
* Able and willing to complete all qualifying diagnostic and functional tests and agrees to comply with study follow-up schedule

Exclusion Criteria:

* Patients with significant organic mitral valve pathology (e.g. myxomatous degeneration, mitral valve prolapse or flail leaflets)
* Myocardial infarction or any percutaneous cardiovascular intervention, cardiovascular surgery, or carotid surgery within 3 months
* Prior surgical, transcatheter, or percutaneous mitral valve replacement
* Untreated clinically significant coronary artery disease (CAD) requiring revascularization
* Hemodynamic instability: Hypotension (systolic pressure <90 mmHg) or requirement for inotropic support or mechanical hemodynamic support
* Any planned cardiac surgery or interventions within the next 6 months (including right heart procedures)
* NYHA class IV (i.e., non-ambulatory)
* Fixed pulmonary artery systolic pressure >70 mmHg
* Severe tricuspid regurgitation
* History of stroke within the prior 3 months or any prior stroke with Modified Rankin Scale ≥ 4 disability
* Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or non-ischemic etiology
* Anatomical pathology or constraints preventing appropriate access/implant of the AccuCinch® Ventricular Repair System (e.g., femoral arteries will not support a 20F system)
* Renal insufficiency (i.e., eGFR of <30ml/min/1.73m2; Stage 4 or 5 CKD)
* Moderate or severe aortic valve stenosis or regurgitation or aortic valve prosthesis
* Fluoroscopic or echocardiographic evidence of severe aortic arch calcification, mobile aortic atheroma, intracardiac mass, thrombus or vegetation
* Active bacterial endocarditis
* Subjects in whom anticoagulation or antiplatelet therapy is contraindicated
* Known allergy to nitinol, polyester, or polyethylene
* Any prior true anaphylactic reaction to contrast agents; defined as known anaphylactoid or other non-anaphylactic allergic reactions to contrast agents that cannot be adequately pre-medicated prior to the index procedure.
* Life expectancy < 1 year due to non-cardiac conditions
* Currently participating in another interventional investigational study
* Implant or revision of any rhythm management device (CRT or CRT-D) prior 3 months or implantable cardioverter defibrillator within the prior 1 month
* Subjects on high dose steroids or immunosuppressant therapy
* Female subjects who are pregnant, of child bearing potential without a documented birth control method, or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2024-01-28 (Actual)

PRIMARY OUTCOMES:
Safety measured by device-related or procedure-related major adverse events (MAEs) | 30-day
  Device-related or procedure-related major adverse events (MAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zapien, MS, CCRA, Study Director — Ancora Heart, Inc.; Kendra Grubb, MD, Principal Investigator — Emory University; Guilherme Silva, MD, Principal Investigator — Baylor St. Luke's Medical Center
Locations (19):
- United States (19):
  - University of California, San Francisco, San Francisco, California
  - Piedmont Heart, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - University of Louisville, Louisville, Kentucky
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Minneapolis Heart Foundation Institute, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mount Sinai, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - PinnacleHealth Cardiovascular Institute, Harrisburg, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Austin Heart, Austin, Texas
  - Baylor College of Medicine St. Luke's Medical Center, Houston, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
  - University of Virginia School of Medicine, Charlottesville, Virginia
  - Virginia Tech Carilion School of Medicine and Research Institute, Roanoke, Virginia
  - University of Washington Medicine, Seattle, Washington